CLINICAL TRIAL: NCT02699775
Title: Effect of 3 Consecutives Botulinum Toxin Injection on Gait Pattern in Stroke Patients
Brief Title: Effect of Repeated Botulinum Toxin Injection on Gait Pattern in Stroke Patients
Acronym: TRITITOX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Collaborators: Fondation Garches (Other)
Responsible Party: Principal Investigator, Nicolas ROCHE, MD PhD, Centre d'Investigation Clinique et Technologique 805
Other Study IDs: 2015-A01671-48
Record Dates: First submitted 2016-03-01; First posted 2016-03-04 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Botulinum Toxins Injection in Stroke Patients
Keywords: Botulinum toxin injections; Stroke; 3D motion analysis; Gait pattern
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic spastic stroke patients: Chronic spastic stroke patients treated regularly with botulinum toxin injection in lower limb muscles
  Interventions: Other: Motion Analysis

INTERVENTIONS:
Other: Motion Analysis — Motion analysis is used to assess the modifications of gait pattern in chronic spastic stroke patients regularly treated with botulinum toxin injection

SUMMARY:
Chronic stroke patients exhibit gait pattern alterations which are mainly due to spasticity and treated with repetitive multifocal botulinum toxin injection(BTI). Several studies demonstrated that single BTI-session in a single muscle of paretic lower limb(LL) improved kinematic gait parameters(GP) but surprisingly none of them assessed the effects of repetitive multifocal BTI on patient's gait pattern and their duration.

The aim was to evaluate the impact of repetitive multifocal BTI-sessions on GP of chronic stroke patients. To that end, gait of patients will be compared using 3D-gait analysis after 3 consecutives BTI sessions.

DETAILED DESCRIPTION:
All the patients will be treated with BTI . These injections will be performed under electrical stimulation control (~5mA). The dose, the number of site of injection per muscle is at the discretion of the physician according to patients' needs and physicians' routine clinical practice. The dilution the most commonly used will be 100 U for 2.5ml (XEOMIN®)

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* a single hemispheric cerebral vascular lesion more than 6 months previously
* able to walk 10 meters without any assistance
* having benefited of at least 2 consecutive BTI sessions, second 3D gait analysis performed at least 3 months after the last BTI.

Exclusion Criteria:

* patient's refusal to participate to the study
* Inability to read the selected text
* Inability to cooperate
* No affiliation to social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: STROKE PATIENTS
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-12-12 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
kinematics gait parameters | 3h
  peak knee flexion in swing phase(°)

SECONDARY OUTCOMES:
spatiotemporal gait parameters | 3h
  Gait velocity (m/s)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas ROCHE, MD PhD, Principal Investigator — Raymond Poincare Hospital
Locations (1):
- Raymond Poincaré hospital, Garches, France

IPD SHARING:
Plan to Share IPD: No